CLINICAL TRIAL: NCT02691169
Title: Comparison of PSMA-based 18F-DCFPyL PET/CT to Conventional Imaging in the Evaluation of Subjects With Castration-Resistant Prostate Cancer
Brief Title: Integrated 18F-labelled PSMA Project
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Katherine Zukotynski, Dr. Katherine Zukotynski, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JNMP-01
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): The subjects will receive the 18F-DCFPyL Injection (less than or equal to 9 mCi (333 MBq)) at visits 2 and 3.
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-DCFPyL is a sterile diagnostic radiopharmaceutical used for PET imaging.

SUMMARY:
There are several new therapies available to treat men with advanced prostate cancer; however, the decision making tools needed to determine the best treatment for these patients are noticeably absent. The prostate-specific membrane antigen (PSMA) is increasingly being recognized as an important target for prostate cancer imaging and determining the most effective therapy. Accordingly, a wide variety of agents are being used to image PSMA. One of these agents is 18F-DCFPyL. In this study the investigators will image men with advanced prostate cancer using 18F-DCFPyL and a positron emission computed tomography (PET/CT) scanner. The investigators will compare the results of 18F-DCFPyL PET/CT for the detection of metastases and monitoring the effects of therapy with conventional imaging (CT, bone scan) and clinical follow-up. In this way, the investigators will evaluate the benefit of using 18F-DCFPyL PET/CT to decide what is the best treatment strategy for a man with advanced prostate cancer.

DETAILED DESCRIPTION:
This is an exploratory single centre, non-randomized, open-label, study in male subjects with metastatic, castrate-resistant PCa (CRPC) being treated with a second-line anti-androgen therapy (enzalutamide or abiraterone). The purpose of the study is to assess if 18F-DCFPyL PET/CT: 1. Shows more sites of metastatic, castrate-resistant PCa (CRPC) compared with standard imaging (bone scan and CT) at baseline and follow-up, 2. Shows response to therapy that is associated with clinical outcome.

This study will image male subjects with CRPC undergoing second-line anti-androgen therapy (enzalutamide or abiraterone) using 18F-DCFPyL PET/CT for detection of metastases and therapeutic monitoring, with correlation to standard-of-care imaging (CT and bone scan) and clinical follow-up over a 1-year time period. Subjects with CRPC and planned treatment with evidence of metastases on standard-of-care imaging (CT and/or bone scan) will undergo a baseline and mid-therapy 18F-DCFPyL PET/CT.

The study design consists of three study clinic visits (screening, baseline 18F-DCFPyL PET/CT, and 8-14 week follow-up 18F-DCFPyL PET/CT) and two follow-up safety phone calls. In addition, all subjects will be followed clinically as per local standard of care with prostate-specific antigen (PSA) blood levels and standard of care imaging for up to one year following the baseline 18F-DCFPyL administration.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years and male
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Subjects starting abiraterone (but naïve to enzalutamide) or starting enzalutamide (but naïve to abiraterone), within approximately 1-7 days of the baseline 18F-DCFPyL PET/CT.
* Prior docetaxel-based chemotherapy is permitted but not required
* Documented metastatic prostate cancer progression as assessed by the treating oncologist with either one or both of the following:

  * Rising PSA over a minimum 1-week interval
  * Radiographic progression in soft tissue and/or bone
* Ongoing androgen deprivation
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Hemoglobin ≥ 90 g/L independent of transfusion
* Platelet count ≥100 x109/L
* Albumin ≥ 30 g/L
* Creatinine < 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min
* Potassium ≥ 3.5 mmol/L

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Abnormal liver functions consisting of any of the following:

  * Total Bilirubin ≥ 1.5 x ULN (except for subjects with documented Gilbert's disease)
  * AST or ALT ≥ 2.5 x ULN (for subjects with known liver metastasis, AST or ALT ≤ 5 x ULN is allowed)
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg)
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 12 months
* Known brain metastasis
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of orally administered hormonal agents.
* Acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a NCI CTCAE (version 4.0) grade of ≤ 1; chemotherapy-induced alopecia and grade 2 peripheral neuropathy are allowed
* Current enrollment in an investigational drug or device study, or participation in such a study within 30 days of the 18F-DCFPyL administration
* Condition or situation which, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Not willing to comply with the procedural requirements of this protocol
* Subjects who have partners of childbearing potential who are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with [F-18]-DCFPyL-related adverse events as assessed by CTCAE v4.0 | Up to 3 days post [F-18]-DCFPyL Injection
  The safety of [F-18]-DCFPyL administration to participants will be assessed by measuring changes from baseline in vital signs (blood pressure, heart rate and oxygen saturation) on the day of injection and through documentation of any other reported adverse events for up to 3 days post-administration.
Extent of baseline disease on [F-18]-DCFPyL imaging compared to extent of baseline disease on conventional imaging in each participant as assessed by counting the total number of lesions on imaging prior to starting hormonal therapy | At the time of initial imaging
  The extent of baseline disease on [F-18]-DCFPyL imaging (total number of lesions) will be compared to the extent of baseline disease on conventional imaging (total number of lesions) to determine [F-18]-DCFPyL imaging sensitivity.

SECONDARY OUTCOMES:
Treatment response on [F-18]-DCFPyL imaging using EORTC criteria will be compared with treatment response on clinical follow-up according to PCWG2 criteria. | 1 year post hormonal therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Zukotynski, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The anonymized individual participant data from this study may be shared with Johns Hopkins University for the purposes of analysis and publication.
Supporting Information: Study Protocol, SAP
Time Frame: October-December 2017